CLINICAL TRIAL: NCT04161261
Title: Minimizing Facial Nerve Stimulation in Cochlear Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Principal Investigator, Sophie McKenny, /Chief Investigator Professor Manohar Bance, Cambridge University Hospitals NHS Foundation Trust
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 272538
Record Dates: First submitted 2019-11-05; First posted 2019-11-13 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Cochlear Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss; Facial Nerve Injury; Nerve Disorders
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Facial Nerve Injuries | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: We will have 2 groups of patients. An Intraoperative group (undergoing cochlear implantation) and a post operative group (with pre existing facial nerve stimulation). The study compares the effectiveness of different pulse shapes within each group, rather than performing a between-group comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IntraOperative Group (Experimental): The intra-operative group consists of patients who have met criteria for cochlear implants. We monitor the facial nerve EMG intraoperatively in all patients, and often get some facial nerve activation when we are testing the implant intraoperatively when we are looking to see if we are getting any hearing nerve responses from electrical stimulation of the implant. We will also measure the facial nerve responses for some other charge-balanced pulse shapes, which are asymmetric and in which either the positive or negative charge is expected to stimulate the nerve. We will only measure these for two electrodes, not for all 12-22 electrodes They will be then invited back post operatively for a second testing during a standard of care visit post switch on for other pulse shapes.
  Interventions: Procedure: Electrical Stimulation
- PostOperative Group (Experimental): The post-operative group, are patients who are actually having facial nerve stimulation on one or more electrodes, and for whom these electrodes are turned down so much they can't hear very well, or are actually turned off because of the facial nerve stimulation. For these patients, we will slowly increase the current levels on the offending electrodes (maximum of two) until they get some facial nerve twitching, and then turn down the current until they do not have stimulation any more. We will do this for all pulse shapes and determine which shape produces the greatest loudness without stimulating the facial nerve. This will be the only testing session for the second group.
  Interventions: Procedure: Electrical Stimulation

INTERVENTIONS:
Procedure: Electrical Stimulation — To measure the facial nerve stimulation threshold for one mid-array and one apical electrode of the implant using the pulse-train stimuli

SUMMARY:
This study aims to understand how to manipulate the electrical stimulation from the cochlear implant to maximize hearing stimulation and minimize facial stimulation. It is know from animal data that the hearing and facial nerves have different sensitivities to things like electrical pulse shape, its pattern, and its duration. It is very unclear however if this applies to human cochlear implant patients, and what the optimal parameters are to selectively stimulate the hearing nerve in humans. The outcomes of this study will be used to more selectively program some patients with severe facial nerve cross stimulation and to inform the development of new types of implant stimulation.

DETAILED DESCRIPTION:
The patients eligible for the study are deaf, and have consented as part of their standard of care to receiving a cochlear implant. There will be no interference with this process in any way. Those patients that are unfortunate to be affected by facial nerve stimulation following receiving their cochlear implant however will be contacted and with the aim to help improve their symptoms as indicated in prior animal studies

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.

  * Male or Female, aged 18 years or above.
  * Unilateral user of a cochlear implant or at least 6 months (post-operative group), or prospective CI user, meeting NICE criteria for implantation (intra-operative group).
  * First language English or sufficiently fluent in English to understand the consenting process
  * Post-lingual onset of severe to profound hearing loss
  * No other handicaps that would interfere with participation in the study in the opinion of the Principal Investigator

Exclusion Criteria:

* Unstable cochlear implant or hearing aid fitting

  * Using medication in an intermittent manner that might influence hearing levels
  * Cognitive or psychological challenges that might lead to variations in attention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2022-05-03 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
To identify stimulus parameters for cochlear implant stimulation that achieve sufficient loudness for hearing, while minimizing stimulation of the facial nerve. | 18 months
  The loudness level, or auditory nerve response at which facial nerve stimulation occurs for different stimulation pulse shapes will be measured for all 24 patients on both groups and help to identify different optimal stimulus parameters.
  By comparing the amount of electrical current required to initiate a facial nerve response for each pulse shape this will determine if there is an optimal type of stimulation to use, to reduce facial nerve stimulation.

SECONDARY OUTCOMES:
To increase scientific understanding of the biology of the auditory and facial nerve's responses to stimulation. | 18 months
  This is a hugely under researched field where we are pioneering techniques and so exact outcome measures may be difficult to quantify in this scientific investigation.
  We are not able to use questionnaires or scientific tools at this stage, however this can be measured through electrical current measurements on the volta software for the Advanced Bionics cochlear implant company.

CONTACTS AND LOCATIONS:
Overall Officials: Manohar L Bance, Professor, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Upon completion of study, data will be disseminated into research community anonymised. IPD will not be accessible to researchers outside the clinical care team.